CLINICAL TRIAL: NCT00796172
Title: Clinic-based Intervention to Improve Medication Adherence to Reduce Cardiovascular Disease Risks
Brief Title: Evaluating the Effectiveness of a Computerized Medication Adherence System at Reducing Cardiovascular Disease Risk Factors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PHCC LP (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, James G. Christian, President, PHCC LP
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 601; R44HL090111 (NIH); 2R44HL090111-02 (NIH)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Cardiovascular Diseases
Keywords: Hypertension; High Blood Pressure; Blood Lipid Management
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

ARMS (2):
- 1 (Experimental): Medication adherence system (MAS) plus counseling from doctors
  Interventions: Behavioral: Medication Adherence System (MAS)
- 2 (Active Comparator): Usual care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Medication Adherence System (MAS) — Participants will receive individualized reports from the MAS and counseling from their doctors. The counseling will focus on adherence to blood pressure and cholesterol management medications.
  Arms: 1
Behavioral: Usual Care — Participants will receive usual care from their doctors and written materials on CVD risk factors.
  Arms: 2

SUMMARY:
High blood pressure and high cholesterol are both causes of cardiovascular disease (CVD), and it is important for people with these conditions to adhere to their medication regimens. This study will evaluate the effectiveness of a computerized program that provides individualized feedback to participants and their doctors for increasing medication adherence among people at risk of developing CVD.

DETAILED DESCRIPTION:
CVD is a disorder that affects the heart's ability to function normally. The most common cause of CVD is narrowing or blockage of the coronary arteries, which supply blood to the heart. There are many risk factors for CVD, including inflammation, high blood pressure, high cholesterol, and obesity. For people who take blood pressure and cholesterol lowering medications, adherence to their medication regimen is another important factor in reducing the risk of CVD. Currently, there are no programs available to assist patients with tracking their medication adherence, despite the fact that non-adherence is a major reason for elevated cholesterol and blood pressure levels. This study will evaluate a computerized medication adherence system (MAS) that provides individualized reports to participants and their doctors with information on identifying and overcoming barriers to medication adherence. The MAS will be evaluated in conjunction with counseling from participants' doctors. The purpose of this study is to evaluate the effectiveness of a computerized MAS plus counseling from doctors for increasing medication adherence and lowering blood pressure and cholesterol levels among people at risk of CVD.

This 1-year study will enroll people with high blood pressure or cholesterol levels who are at risk of CVD. At a baseline study visit, participants will undergo blood pressure measurements, a blood collection, and a medication review. Participants will be randomly assigned to either the MAS group or a usual care group. Participants in the MAS group will use the computerized MAS program and answer questions about their medication regimens. Reports will then be generated for both the participants and their doctors. Participants will meet with their doctors to review the reports and discuss their medications and CVD risks. Participants in the usual care group will receive written materials on CVD risk factors, and they will receive usual care from their doctors. At a 6-month visit, participants in the MAS group will undergo a medication review, blood pressure measurements, and interviews with study staff. They will also enter their medication information into the MAS and meet with their doctors to discuss the generated report. Participants in the usual care group will not take part in any study procedures at 6 months. At a 12-month visit, all participants will undergo blood pressure measurements, a blood collection, and a medication review. Participants in the MAS group will also complete questionnaires to assess the usefulness of the MAS computer program.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed one or more antihypertensive and/or lipid management medications
* Living independently
* Has a literacy level that will enable them to successfully navigate the MAS and read associated reports (i.e., approximately a sixth grade reading level)

Exclusion Criteria:

* Current substance use or abuse
* Recent (in the 6 months before study entry) heart attack, stroke, peripheral vascular disease, or other medical condition that limits a potential participant's ability to complete the necessary visits to the outpatient clinic site, to use the MAS, and to complete study assessments
* Residing in assisted living or a nursing home situation
* Medical condition for which survival is expected to be unlikely in the 1 year after study entry
* Unable to read or use a computer with a computer mouse

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Medication adherence and associated changes in blood pressure and lipid profiles | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: James G. Christian, MSW, MABS, Principal Investigator — PHCC LP
Locations (1):
- PHCC LP, Pueblo, Colorado, United States